CLINICAL TRIAL: NCT04937335
Title: Clinical Features and Risk Factors of Craniopharyngioma With Tumoral Hemorrhage
Brief Title: Craniopharyngioma With Tumoral Hemorrhage
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Kai Shu, Prof. Dr., Tongji Hospital
Other Study IDs: kaishu1
Record Dates: First submitted 2021-06-07; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Craniopharyngioma; Apoplexy
Keywords: craniopharyngioma; endocrine; risk factor; tumoral hemorrhage
MeSH Terms: conditions — Craniopharyngioma; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-hemorrhage group: Patients recognized as craniopharyngioma pathologically without tumoral hemorrhage observed during the operation
- Hemorrhage group: Patients recognized as craniopharyngioma pathologically with tumoral hemorrhage observed during the operation
  Interventions: Other: intratumoral hemorrhage

INTERVENTIONS:
Other: intratumoral hemorrhage — Patients who were recognized as craniopharyngioma pathologically with tumoral hemorrhage observed during the operation were enrolled in the hemorrhage group.
  Groups: Hemorrhage group

SUMMARY:
Clinical data of 185 consecutive patients receiving resective operation with a pathological diagnosis of craniopharyngioma in our hospital between January 2013 and February 2021 were collected. Among these patients, 18 of them were recognized as craniopharyngioma with tumoral hemorrhage during the operation.

DETAILED DESCRIPTION:
For each case, age, gender, smoking status, alcohol intake, past history, symptoms, blood pressure, blood cell count, blood biochemical tests, coagulation tests, hormone tests, radiological results, surgical treatment and the outcome at discharge were collected. The first test result after admission and before the operation was taken for the items of blood tests with multiple times in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* receive resective operation with a pathological diagnosis of craniopharyngioma in our hospital
* enter our hospital between January 2013 and February 2021

Exclusion Criteria:

* have a non-craniopharyngioma or unverified pathological diagnosis at discharge
* have received surgical or radiological treatment on the sellar region
* receive treatment of coagulation modulation, immunosuppressive agents or chemotherapeutic drugs
* combine with other clinical emergencies including acute myocardial infarction, cerebral stroke, trauma and sepsis at admission
* have been diagnosed with other tumors, hematological diseases, autoimmune diseases, liver failure or renal failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with a pathological diagnosis of craniopharyngioma
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
craniopharyngioma with tumoral hemorrhage | during the operation
  Current study is a case-control study whose primary outcome is tumoral hemorrhage observed during the operation, which devided the craniopharyngioma patients into hemorrhage group and non-hemorrhage group.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Shu, MD, Study Director — Tongji Hospital

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the questions asked in this study, survey respondents were assured raw data would remain confidential and would not be shared.